CLINICAL TRIAL: NCT04436666
Title: The Effect of Virtual Reality and Ice Application on Fear of Self-injection and Self-test, Pain and State Anxiety Levels in Patients With Type 2 Diabetes
Brief Title: Virtual Reality, Ice Application and Self-injection and Self-test Fair, Pain and State Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, seher ÇEVİK, Principal Investigator, Inonu University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: seher cevik
Record Dates: First submitted 2020-06-15; First posted 2020-06-18 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Injection Site Irritation; Fear of Pain
Keywords: Insulin injection; fear of injection; Ice application; Virtual reality
MeSH Terms: conditions — Iatrophobia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ice Application (Experimental): Music-funded, park, nature and seaside walks, submarine, museum, with virtual reality glasses (Bobo VR Z4 Binocular Glasses and 5.7 inch 1440x2560 pixel display resolution, China) for 10 minutes to diabetic patients before blood glucose measurement and insulin injection The videos that the patient wants to watch will be watched from videos such as his trip Studies have indicated that these videos are relaxing environments, and motion videos should not be watched to reduce nausea and vomiting.
  Interventions: Other: Ice Application
- Virtual Reality (Experimental): Before the blood glucose measurement and insulin injection, patients with diabetes will be given ice for 5 minutes. It is planned to apply ice cubes in liquid-proof ice bags.
  Interventions: Device: motivational video production through virtual reality glasses
- control (No Intervention): No Intervention

INTERVENTIONS:
Device: motivational video production through virtual reality glasses — Music-funded, park, nature and seaside walks, submarine, museum, with virtual reality glasses (Bobo VR Z4 Binocular Glasses and 5.7 inch 1440x2560 pixel display resolution, China) for 10 minutes to diabetic patients before blood glucose measurement and insulin injection The videos that the patient wants to watch will be watched from videos such as his trip Studies have indicated that these videos are relaxing environments, and motion videos should not be watched to reduce nausea and vomiting.
  Arms: Virtual Reality
Other: Ice Application — Before the blood glucose measurement and insulin injection, patients with diabetes will be given ice for 5 minutes. It is planned to apply ice cubes in liquid-proof ice bags.
  Arms: Ice Application

SUMMARY:
AİM:The aim of this study is to control the fears and anxieties of Type 2 diabetics in insulin injection and blood glucose measurement with motivational videos and Ice applications to be applied with virtual reality glasses.

Material and Methods: The research is designed as a semi-experimental model with pretest-posttest control groups. The research will be carried out in the endocrine services located in Turgut Özal Medical Center in Malatya province. The universe of the research will be 2113 Type 2 diabetes patients who are being treated in the hospital specified on the specified dates, who are injecting insulin and following blood sugar. According to the analysis of the power, the sample of the research is composed of an experiment effect of 0.5% with bilateral significance level, 95% confidence interval determined with 5% error level, the experiment group to be applied with 80% Reality with 80% representation power, and the control group with 80 ice application. will create a total of 240 Type 2 diabetes patients.In the collection of the data, the Participant Presentation Form developed by the researcher, Diabetes Fear of Self Injecting and Self-testing Questionnaire-D-FISQ, State Anxiety Scale and VAS will be used.

DETAILED DESCRIPTION:
VR is a relatively new human-computer interaction tool in which a person becomes an active participant in a virtual world. Sensory cues of VR, especially the precise control of auditory, tactile and olfactory systems, enhances the reality of the virtual environment. As a result, users feel that they can look around and enter the simulated environment. The virtual environment provides sensory information such as visual, auditory, movement, virtual or artificial, and makes the individual feel similar to real life.

Ice application has been used as a topical pain reliever for centuries. It works through a variety of mechanisms, such as slowing the transmission of peripheral nerve fibers, promoting sensory competition, and reducing the release of inflammatory and nociceptive mediators. Ice application is cheap, easily accessible and reaches its purpose relatively quickly to skin anesthesia. Apart from these effects, it also reduces pain by activating the Door-Control mechanism, stimulating the touch receptors and increasing the release of endogenous opioids.

ELIGIBILITY:
Inclusion Criteria:

* Being literate,
* Injecting insulin at least twice a day,
* Following blood sugar at least twice a day,

Exclusion Criteria:

* Having any psychiatric diagnosis,

  * communication barriers
  * The patient has any diagnosis, such as epilepsy, that will trigger seizures.
  * Any diagnosis, such as vertigo, that causes dizziness in the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Injection fear reduction | 1 month
  (Diabetes Fear of Self Injecting and Self-testing Questionnaire-D-FISQ) D-FISQ was developed by Snoek et al. (1997) to measure the fear of self-injection and testing in individuals with diabetes who need insulin. D-FISQ with 15 expressions consists of two sub-dimensions, fear of self-injecting-FSI, 6 expressions, and fear of self-testing (FST, 9 expressions). Each statement has a 4-point Likert-type rating ranging from 1 to 4 (1 = almost never, 2 = sometimes, 3 = often, 4 = almost always). The evaluation of the inquiry form can be done by taking the average or raw score for the two sub-dimensions and the whole form. As the scores obtained from the scale increase, fear levels increase. Internal consistency coefficient of the scale is 0.96.
anxiety reducation | 1 month
  State Anxiety Scale The scale, which was developed by Spielberger et al in 1970, was adapted to Turkish by Öner and LeCompte (1974). The emotions or behaviors expressed in the scale items are answered by marking one of the options such as (1) none, (2) a little, (3) a lot, and (4) completely. The scale containing twenty expressions contains 10 inverse (1, 2, 5, 8, 10, 11, 15, 16, 19, 20) expressions. While the reverse expressions expressing positive emotions are scored, those in one weight degree are converted into four, and those in four weight degrees into one. In the scoring, the total weighted score of the inverse statements is subtracted from the total weighted score and 50, an unchanged value, is added to this number. The total score value obtained from the scale can range from 20 to 80 points. A high score indicates that the level of anxiety is high. The total score value is evaluated as 20-39 mild anxiety, 40-59 moderate anxiety, and 60-79 severe anxiety.
pain relief | 1 month
  (Visual Analogue Scale -VAS) This scale, which is used to measure subjectively perceived pain, was developed by Price et al. (1983), and has been used in many studies to evaluate the intensity of pain, it has been found to be reliable and valid. It is a 10 cm scale with "painlessness" on one end and "severe pain" on the other. Individuals participating in the study are asked to mark the level of pain severity they feel at the moment, explaining that the number "0" on the scale means that I do not feel any pain and the pain intensity increases as the numbers grow and the number "10" means the most severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: seher ÇEVİK, Principal Investigator — Inonu University
Locations (1):
- seher ÇEVİK, Malatya, Turkey (Türkiye)

REFERENCES:
- [Background] Cevik S, Yagmur Y. Impact of intolerance of uncertainty on psychological well-being in pregnant women with or without miscarriage risk. Perspect Psychiatr Care. 2018 Jul;54(3):436-440. doi: 10.1111/ppc.12297. Epub 2018 May 25. PMID 29799614